CLINICAL TRIAL: NCT02074891
Title: Sustainable Healthcenter Implementation PrEP Pilot Study
Acronym: SHIPP
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: CDC Foundation (Other); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Karen Hoover, Lead, Prevention Research Team, Centers for Disease Control and Prevention
Other Study IDs: CDC-NCHHSTP-6511
Record Dates: First submitted 2014-02-24; First posted 2014-02-28 (Estimated); Last update posted 2024-05-28 (Actual); Status verified 2016-02

CONDITIONS: HIV Chemoprophylaxis; HIV Preexposure Prophylaxis
Keywords: preexposure prophylaxis; PrEP; HIV
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Tenofovir; Racivir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dried blood spots
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Persons prescribed PrEP: adults prescribed daily oral antiretroviral preexposure prophylaxis (PrEP) with the coformulated TDF/FTC to reduce HIV acquisition.
  Interventions: Drug: coformulated TDF/FTC

INTERVENTIONS:
Drug: coformulated TDF/FTC — Daily oral dose of coformulated TDF/FTC
  Other Names: Truvada; Tenofovir disoproxil fumarate (TDF); Emtracitabine (FTC)

SUMMARY:
A health services implementation pilot study, conducted with an observational cohort of HIV-uninfected persons including men who have sex with men, heterosexual women and men, and injection drug users receiving daily oral antiretroviral preexposure prophylaxis (PrEP) at four federally qualified health centers that provide sexual health and primary care services to communities with high HIV incidence/prevalence.

ELIGIBILITY:
Inclusion Criteria:

* adult
* documented without HIV infection (acute or established)
* report sexual behaviors that indicate substantial risk of HIV acquisition
* report injection-related behaviors that indicate substantial risk of HIV acquisition

Exclusion Criteria:

* <18 years of age
* documented HIV infection (acute or established)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1200 adult men who have sex with men, injection drug users, and heterosexually-active men and women who are at substantial risk of acquiring HIV infection and initiate the use of daily oral antiretroviral preexposure prophylaxis (PrEP) with TDF/FTC
Sampling Method: Non-Probability Sample
Enrollment: 1420 (Actual)
Dates: Start 2014-10; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Clinical safety | Every 3 months up to 36 months
  Side effects, rates of renal adverse events, rates of atraumatic bone fractures, HIV infections with/without virus with mutations associated with TDF or FTC resistance, documented at clinical visits while prescribed PrEP
Medication adherence | Every 3 months up to 36 months
  Self-reported medication adherence and detection of tenofovir in dried blood spots at each clinical visit while prescribed PrEP
Behavioral Responses | Every 3 months up to 36 months
  Trends in sexual and injection HIV acquisition risk behaviors among patients measured at each clinic visit while prescribed PrEP

SECONDARY OUTCOMES:
Costs | Up to 3 years
  Source of payment, cost, and reimbusement for medication and clinical care associated with each clinical visit for PrEP
Clinical practice variation | Every 3 months up to 36 months
  Variation in clinical practices at each clinic visit for PrEP-related care relative to PHS PrEP guidelines, and the relationship of clinical practices to patient outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Dawn K Smith, MD, MS, MPH, Study Chair — Centers for Disease Control and Prevention; Rebecca Cook, MPH, Study Director — CDC Foundation
Locations (5):
- United States (5):
  - Whitman Walker Health, Washington D.C., District of Columbia
  - Access Community Health Network - Grand Boulevard Health and Specialty Center, Chicago, Illinois
  - Howard Brown Community Health Center, Chicago, Illinois
  - Open Arms Healthcare Center, Jackson, Mississippi
  - Strawberry Mansion Health Center, Philadelphia, Pennsylvania